CLINICAL TRIAL: NCT04401449
Title: Cardiopulmonary Inflammation and Multi-System Imaging During the Clinical Course of COVID-19 Infection in Asymptomatic and Symptomatic Persons (COVID ARC 19)
Brief Title: Cardiopulmonary Inflammation and Multi-System Imaging During the Clinical Course of COVID-19 Infection in Asymptomatic and Symptomatic Persons
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 200113; 20-CC-0113
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11-19

CONDITIONS: Acute and Long Term Effects of COVID-19 on Systemic Inflammation; Acute and Long Term Effects of COVID-19 on Lung Function; Acute and Long Term Effects of COVID-19 on Cardiac Function; Acute and Long Term Effects of COVID-19 on Kidney Function; Acute and Long Term Effects of COVID-19 on Brain Function
Keywords: Immunological Function; SARSCoV-2; Neurologic Function; Cardiac Function; Pulmonary Function; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acutely illl subjects: COVID-19 subjects treated at the Clinical Center, followed through recovery and into convalescence
- Recovered subjects: COVID-19 subjects who were treated at other hospitals, followed through recovery and into convalescence

SUMMARY:
Background:

COVID-19 virus infection differs among people. Some people have no or mild symptoms. For others, COVID-19 is life threatening and causes damage to the body s organs. Researchers want to better understand the virus to learn how to kill it.

Objective:

To understand how the COVID-19 virus causes wide differences in how sick one can become from the infection.

Eligibility:

People ages 18-80 with COVID-19 infection

Design:

Participants will be screened with a review of their medical records.

Participants who enter the study at the beginning of their COVID-19 infection will stay in the hospital until they are healthy enough to go home. Those who enter after they have recovered may need to stay in the hospital 1-2 nights to perform the study tests.

Participants will have MRI and CT scans of the brain, heart, and lungs. They will lie in a machine that takes pictures of the body. For the MRI, soft padding or a coil will be placed around their head and chest. They may receive a dye injected into a vein.

Participants will have an ultrasound of the kidneys and heart.

Participants will provide blood and urine samples. They will provide nasal swabs.

Participants will have a bronchoscopy. A thin tube will be placed through the nose or mouth into the airway. Saltwater will be squirted into the lungs and removed by suction.

Participants may provide a spinal fluid sample. A needle injected into the spinal canal will obtain fluid.

Participants will have lung and heart function tests.

At various points after recovery, participants will repeat many of these tests.

DETAILED DESCRIPTION:
Study Description: This protocol will enroll patients within a 50 mile radius of Bethesda, Maryland, to the Clinical Center in a longitudinal study using granular clinical observations including pulmonary and cardiac functional assessments, comprehensive immunologic evaluations, and innovative imaging. Sequential analysis of blood, bronchoalveolar lavage, and spinal fluid, with simultaneous serial imaging can provide insights into mechanisms associated with the initiation, progression and resolution of organ dysfunction and systemic inflammation due to COVID-19 infection.

Objectives:

Primary objective:

To link inflammatory responses present in blood, bronchoalveolar lavage, spinal fluid, and with imaging of COVID-19 target organs (lungs, heart and brain) during the earliest stages of infection and at subsequent time points as the infection and host responses evolve, through recovery.

Secondary objectives

Assess the long-term effects of COVID-19 infection on immunologic, neurologic, cardiac and pulmonary function

Endpoints:

1. Measure inflammatory responses present in blood, bronchoalveolar lavage, and spinal fluid during the course of COVID-19 infection
2. Obtain imaging of target organs during the course of COVID-19 infection
3. Evaluate long-term effects of COVID-19 infection on immunologic, cardiac, pulmonary and neural function

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

Subjects within 1-28 days of documented COVID-19 infection for acute care:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 to 80 years

  * Only a minority of children and adolescents have been described as developing serious illness with COVID-19 infection. As such, this is not an age group at significant risk from complications due to this infection. Adults older than 80 years of age represent a group with the greatest risk of mortality from COVID-19 infection. The presence of significant co-morbidities requiring care that cannot be

provided at the CC would present a disadvantage to them to have their acute care provided for in the CC.

* Documentation of positive SARSCoV-19 test by nucleic acid detection (COVID-19 infection , RT-PCR)
* Ability of subject to understand and the willingness to sign a written informed consent document.

Subjects during recovery phase of the acute illness (day 28 +/- 7 days to 12 weeks) and convalescent phase (Week 13 up to 12 months), Year 2 convalescent phase (13 24 months), Year 3 convalescent phase (25 36 months) after recovery if care has been received at a facility outside of NIH:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged 18 to 80 years.
* Study participants will be invited to continue their participation in the study in years 2 and 3 based on the results of their tests from the first year and their willingness to continue for the two additional years. If test results of imaging, blood, pulmonary function and or bronchoscopy have returned to normal at the end of one year, the need for further cardiopulmonary testing will be assessed for each patient. Anyone who is invited to continue in the 2nd and 3rd years may discontinue their participation at any time.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnancy or lactation Study participants who are enrolled in the study and become pregnant during the enrollment period will be discontinued from further study participation. Exposure to radiation or radiographic contrast agents for research purposes .only would not be warranted for a pregnant woman and her fetus.
* Serious mental illness (e.g. schizophrenia, manic depression) that would limit the ability of the participant to participate willingly into the study.

  -- The conduct of the study requires participation in studies that may be unduly stressful (e.g. MRI, bronchoscopy).
* Severe claustrophobia that would prohibit the conduct of imaging by MRI even if sedation is provided.
* Cardiac pacemaker or implantable defibrillator unless it is safe for MRI
* Cerebral aneurysm clip unless it is safe for MRI
* Brain stimulator (e.g. TENS-Unit) unless it is safe for MRI
* Any type of ear implant unless it is safe for MRI
* Foreign body in the eye (e.g. metal shavings)
* Metal shrapnel or bullet
* Any implanted device (e.g. insulin pump, drug infusion device
* Patients requiring mechanical ventilation at an outside hospital prior to transfer. Transporting these patients adds risk to their care.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men or women, 18 - 80 years of age, a) within 1- 28 days (+/- 7 days) of documented COVID-19 infection for acute care (n=150) with subsequent follow-up during recovery (28 +/- 7 days to 12 weeks) and then during convalescence (Week 13 to 12 months - year 1), year 2 convalesecent phase and year 3 convalesecent phase. Each Phase visit can be done out of window as per PI discretion. OR b) if care for acute COVID-19 infections was given at an outside site, participants would be evaluated during recovery (28 +/- 7 days to 12 weeks, during convalescence (Week 13 to 12 months - year 1), year 2 - convalesecent phase and year 3 - convalesecent phase) Each Phase visit can be done out of window as per PI discretion.
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Inflammatory responses of cells in lung and circulation | From onset of illness in hospital through acute phase ( days 1 28 more or less 7
  Link inflammatory responses present in blood and bronchoalveolar lavage with imaging of COVID-19 target organs (lungs, heart, brain ) during the earliest stages of infection and at subsequent time points as the infection and host responses evolve, through recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F Suffredini, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (2):
- United States (2):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided
The protocol is silent about Individual Participant Data (IPD) sharing.

REFERENCES:
- [Background] Mao L, Jin H, Wang M, Hu Y, Chen S, He Q, Chang J, Hong C, Zhou Y, Wang D, Miao X, Li Y, Hu B. Neurologic Manifestations of Hospitalized Patients With Coronavirus Disease 2019 in Wuhan, China. JAMA Neurol. 2020 Jun 1;77(6):683-690. doi: 10.1001/jamaneurol.2020.1127. PMID 32275288
- [Background] Driggin E, Madhavan MV, Bikdeli B, Chuich T, Laracy J, Biondi-Zoccai G, Brown TS, Der Nigoghossian C, Zidar DA, Haythe J, Brodie D, Beckman JA, Kirtane AJ, Stone GW, Krumholz HM, Parikh SA. Cardiovascular Considerations for Patients, Health Care Workers, and Health Systems During the COVID-19 Pandemic. J Am Coll Cardiol. 2020 May 12;75(18):2352-2371. doi: 10.1016/j.jacc.2020.03.031. Epub 2020 Mar 19. PMID 32201335
- [Derived] Huapaya JA, Higgins J, Kanth S, Demirkale CY, Gairhe S, Aboye EA, Regenold D, Sahagun SJ, Pastor G, Swaim D, Dewar R, Rehman T, Highbarger HC, Lallemand P, Laverdure S, Adelsberger J, Rupert A, Li W, Krack J, Teferi G, Kuruppu J, Strich JR, Davey R, Childs R, Chertow D, Kovacs JA, Barnett C, Torabi-Parizi P, Suffredini AF; COVID-ARC Study Group. Vaccination Ameliorates Cellular Inflammatory Responses in SARS-CoV-2 Breakthrough Infections. J Infect Dis. 2023 Jun 28;228(1):46-58. doi: 10.1093/infdis/jiad045. PMID 36801946
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-CC-0113.html